CLINICAL TRIAL: NCT01528423
Title: Evaluation of the XtremeCT Device for the Assessment of Bone
Acronym: XtremeCT
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH15265
Record Dates: First submitted 2012-01-25; First posted 2012-02-08 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Peripheral Bone Density
Keywords: XtremeCT; Density; pQCT; Turnover; Bone; short-term reproducibility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples taken for measurement of PINP, CTX, PTH, calcium, creatinine, albumin, testosterone, IGF-1, IGFBP-3 and SHBG
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Men 16 - 18yrs
  Interventions: Procedure: XtremeCT
- Men 30 - 32 yrs
  Interventions: Procedure: XtremeCT
- Men 70 yrs +
  Interventions: Procedure: XtremeCT
- Women 16 - 18 yrs
  Interventions: Procedure: XtremeCT
- Women 30 - 32 yrs
  Interventions: Procedure: XtremeCT
- Women 70 yrs +
  Interventions: Procedure: XtremeCT

INTERVENTIONS:
Procedure: XtremeCT — The scanning protocol for each subject will be as follows: Non-dominant, non-fractured distal radius x 2 with repositioning between scans Non-dominant, non-fractured distal tibia x 2 with repositioning between scans using XtremeCT device and Non-dominant forearm x 2 with repositioning between scans Non-dominant lower leg x 2 with repositioning between scans using standard pQCT device
  Other Names: Device: XTremeCT; Device: pQCT

SUMMARY:
The research is intended to evaluate the short-term reproducibility of the XtremeCT device for measurements of peripheral bone density and bone structure in population-based volunteers from different age groups and to compare the XtremeCT with current peripheral quantitative computed tomography (pQCT) technology. The investigators will also assess the correlation between XtremeCT measurements of bone structure with hormones and biochemical markers of bone turnover.

DETAILED DESCRIPTION:
The investigators plan to perform high resolution-peripheral quantitative computer tomography (HR-pQCT) using the XtremeCT device in future research studies to investigate the structural changes that occur during adolescence and young adulthood to attain peak bone mass (peak bone strength) and to evaluate the structural effects of anabolic treatments for osteoporosis. This preliminary study will establish the short term precision of the device in the populations that the investigators are likely to study and whether the new device is superior to their current pQCT device. It will also provide information on how measurements from the new device relate to bone turnover markers, which are one of their standard assessments of bone metabolism. They will also determine whether hormones that influence bone metabolism have specific effect on different components of bone structure. By providing data on the size and variability of differences in bone structure by gender and at important stages of skeletal development (end of longitudinal growth, peak bone mass and aging) this study will also form the basis of power calculations for future longitudinal studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Willing to participate
* Aged 16-18, 30-32 or ≥ 70 years

Exclusion Criteria:

* Unable to give informed consent
* Prior fracture of both wrists or both tibiae
* Confirmed fracture of three or more vertebrae between the levels of L1 and L4, or degenerative bone disease preventing three or more vertebrae from being evaluated
* Diagnosis of any disease or condition known to affect bone metabolism
* Use of any medication known to affect bone metabolism
* Pregnancy

  * 16-18 and 30-32 year old women will undergo a urine-based pregnancy test at the study site prior to undergoing any study procedures to avoid unnecessary exposure of a foetus to ionizing radiation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To calculate the short-term reproducibility of the XtremeCT device for measurements of bone density and bone structure at the distal radius and tibia in a) teenagers, b) young adults and c) older adults | Data will be analysed following completion of scans. Participants are only involved for 1 day.

SECONDARY OUTCOMES:
A secondary endpoint will be agreement between HR-pQCT and pQCT measurements made in the same individuals and at the same measurement sites using the XtremeCT and XCT-2000 respectively | Data will be analysed following completion of scans. Participants are only involved for 1 day.
A secondary endpoint will be correlation of bone turnover markers with XtremeCT measurements | Data will be analysed following completion of scans. Participants are only involved for 1 day.
A secondary endpoint will be correlation of hormones with XtremeCT measurements | Data will be analysed following completion of scans. Participants are only involved for 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorks, United Kingdom